CLINICAL TRIAL: NCT04395547
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Study to Investigate the Safety and Efficacy of JointAlive™ on Improving Knee Joint Function in Adults With Mild to Moderate Knee Osteoarthritis
Brief Title: Safety and Efficacy of JointAlive™ on the Knee-joint Function in Adults With Knee Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chenland Nutritionals Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20GJHC
Record Dates: First submitted 2020-05-13; First posted 2020-05-20 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- JointAlive™ (Experimental)
  Interventions: Dietary Supplement: JointAlive™

INTERVENTIONS:
Dietary Supplement: JointAlive™ — Combination herbal extract
  Arms: JointAlive™
Dietary Supplement: Placebo — Combination placebo product
  Arms: Placebo

SUMMARY:
Osteoarthritis (OA) is a joint disorder caused by wear and tear on the joint over time; as a result, the protective cartilage of the bone in the joint gradually wears down. The lifetime risk of developing OA in the knee, with symptoms such as pain, aching, and stiffness, is 40% in men and 47% in women. It is estimated that approximately 19% of Americans aged 45 and older are affected by knee OA. Knee OA accounts for 83% of the global burden caused by all OA types. Pain and stiffness in knees, a large weight-bearing joint, often leads to disability, which interferes with daily life activities and demands expensive medical treatments or care. Due to the limitations of current OA treatment methods, there is an increasing demand for effective and safer alternatives, such as natural health products with pain-relieving potential. The investigational product, JointAlive™, is a supplement designed to alleviate knee OA symptoms and to improve knee functionality. The present study will investigate the safety and efficacy of JointAlive™ in reducing knee OA symptoms and improving joint functionality in an otherwise healthy adult population with mild to moderate knee OA. JointAlive™ is a proprietary blend of Epimedium brevicornum Maxim leaves, Dioscorea nipponica Makino rhizome, Salvia miltoiorrhiza Bunge root and rhizome extracts

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a joint disorder caused by wear and tear on the joint over time; as a result, the protective cartilage of the bone in the joint gradually wears down. The lifetime risk of developing OA in the knee, with symptoms such as pain, aching, and stiffness, is 40% in men and 47% in women. It is estimated that approximately 19% of Americans aged 45 and older are affected by knee OA. Knee OA accounts for 83% of the global burden caused by all OA types. Pain and stiffness in knees, a large weight-bearing joint, often leads to disability, which interferes with daily life activities and demands expensive medical treatments or care. Losina et al. reported that in the United States, the average lifetime costs for symptomatic knee OA management is $12,400 USD, but the cost can be higher with knee surgeries for advanced OA. The economic burden is expected to continue increasing in the near future due to the aging population and increasing prevalence of obesity in many developed countries.

Although the exact etiology of OA is unknown, many risk factors are associated with the development of knee OA, such as obesity, repetitive use of joints, age, and previous knee injury or surgery. Multiple studies have shown a positive association between pro-inflammatory cytokines (e.g. tumor necrosis factor (TNF)-α, interleukin (IL)-1β, and IL-6) and OA development. Cytokine-induced nuclear factor-κB (NF-κB) activation can stimulate articular chondrocyte catabolism and extracellular matrix degradation, leading to the breakdown of articular cartilage. The severity of cartilage disintegration and osteophyte (a bony outgrowth) formation can be identified radiographically and used for the Kellgren-Lawrence (KL) grading scheme. A KL score of one (doubtful narrowing of the joint space with possible osteophyte formation) is considered possible OA, while a score of two (possible narrowing of joint space with definite osteophyte formation) or three (definite narrowing of joint space and moderate osteophyte formation) is considered as a definite/mild OA.

It is crucial to treat OA early, before it develops into more severe cases and causes mobility disability. The first step of OA treatment is exercise and/or physiotherapy, which has demonstrated long-term benefits but often difficult to maintain compliance. Once the pain is difficult to manage, over-the-counter medicines such as Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) are introduced to provide relief. NSAIDs are effective in reducing pain, however, long-term usage requires medical supervision. Chronic NSAID use is associated with high incidence of adverse events such as upper gastrointestinal tract problems, kidney and liver injury, hypertension, and congestive heart failure. When the abovementioned treatments are ineffective, intra-articular injections of hyaluronic acid, cortisol, or platelet rich plasma are applied and proven effective, but they can be costly and may cause reactive flares or infections at the injection site. Surgery serves as last resort; it is a successful treatment for advanced OA, but it is invasive and may increase risks of infection, bleeding, and deep vein thrombosis. Given the limitations of current OA treatment methods, there is an increasing demand for effective and safer alternatives, such as natural health products with pain-relieving potential.

The investigational product, JointAlive™, is a supplement designed to alleviate knee OA symptoms and to improve knee functionality. JointAlive™ contains extract from flowering plants that are endemic to China.The main bioactive component is icariin; a flavonoid glycoside demonstrating various antioxidant and anti-inflammatory benefits. Numerous in vitro cell culture studies showed that icariin has the potential to suppress inflammatory pathways involved in OA. In rodent OA models, joint injection of icariin for 32 and 84 days was found to protect the articular cartilage from degeneration.

The present study will investigate the safety and efficacy of JointAlive™ in reducing knee OA symptoms and improving joint functionality in an otherwise healthy adult population with mild to moderate knee OA. Based on the previous studies conducted on the ingredients of this investigational product and their previous application in OA, participants identifying mild or moderate OA in a target knee will be investigated in this study. As OA is a secondary complication in sports injuries as well as a primary development during aging, an age range between 40-75 years will be considered for enrolment. The Kellgren-Lawrence grading scale will be used to confirm OA. As well, BMI cut offs between 18.5 and 29.9 kg/m2 will be considered to excluded those with complications due to obesity and the associated increase in concomitant medication use. To allow for pain relief, as this study involves a placebo group, a rescue medication will be provided. However, in order to ensure that the capture of pain in the target knee is unbiased, participants will be required to abstain from the rescue medication use for 48 hours prior to their clinic visits. Confounders due to medical history and concomitant medications will be ensured by several targeted exclusion criteria with the intent of decreasing potential confounders of the study results.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 40 and 75 years of age, inclusive
2. BMI between 18.5 to 29.9 kg/m2, inclusive
3. Female participant is not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening Or,

   Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
4. Self-reported pain or swelling in target knee
5. The diagnosis of mild to moderate osteoarthritis as confirmed by the Qualified Investigator using qualifiers based on physical exam, medical history and x-ray report qualified as mild to moderate by the radiologist
6. Agrees to refrain from taking any pain relievers during the study, except acetaminophen as a rescue medication specified by the study site
7. Agrees to refrain from taking rescue medication for 48 hours prior to study visits
8. Agrees to maintain current diet and current exercise routine throughout the study
9. Willingness to complete questionnaires, records, and diaries associated with the study and to complete all clinic visits
10. Provided voluntary, written, informed consent to participate in the study
11. Healthy as determined by medical history, laboratory results, and physical exam as assessed by the Qualified Investigator (QI)

Exclusion Criteria:

1. Allergy, sensitivity, or intolerance to the investigational product's active or inactive ingredients
2. Allergy to rescue medication
3. Women who are pregnant, breast feeding, or planning to become pregnant during the study
4. Clinically significant abnormal laboratory results at baseline as assessed by the QI
5. Individuals who are unable to give informed consent
6. Injury in the target knee within the past 3 months
7. Intraarticular injections in the target knee within the past 6 months, or plan to have intraarticular injections during the study
8. Individuals with knee joint diseases, such as rheumatoid arthritis, gouty arthritis, septic arthritis or any other infective arthritis
9. Self-reported history of gout or pseudo gout within the past 6 months
10. Skin defects (e.g. skin and soft tissue infections that cause necrosis of the skin, or post-burn contractures) and ulcers around the affected knee joint, as assessed by the QI
11. History of knee surgery or replacement in the target knee, or any non-knee surgical procedures that may impact the study outcomes as assessed by the QI
12. Individuals with muscle or skeletal disorders as assessed by the QI
13. Unstable metabolic disease or chronic diseases as assessed by the QI
14. In a state of acute exacerbation or seizure of chronic disease
15. Type I or Type II diabetes
16. History of or current diagnosis with severe cardiopulmonary, kidney and/or liver dysfunctions, with the exception of history of kidney stones in participants who are symptom free for 6 months
17. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
18. Current or history of any significant diseases of the gastrointestinal tract including diarrhea or dysentery as assessed by the QI
19. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
20. Self-reported confirmation of medical or neuropsychological condition and/or cognitive impairment that, in the QI's opinion, could interfere with study participation
21. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
22. Verbal confirmation of blood/bleeding disorders as assessed by the QI
23. Individuals with an acute infectious disease, autoimmune disease or are immune-compromised
24. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis
25. Current use of prescribed medications listed above
26. Current use of over-the-counter medications, supplements, foods and/or drinks listed above
27. Use of medical cannabinoid products
28. Chronic use of cannabinoid products (>2 times/week) and is unwilling to stop use for the duration of the study. Occasional use to be assessed by the QI on a case-by-case basis
29. Alcohol or drug abuse within the last 12 months
30. High alcohol intake (average of >2 standard drinks per day)
31. Blood donation 30 days prior to screening, during the study, or a planned donation within 30 days of the last study visit
32. Participation in other clinical research studies 30 days prior to screening
33. Any other condition, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Participants on the following concurrent prescribed medications and/or treatments will be excluded during enrollment unless they have been taken off these therapies by their family physician. In the latter event, the frequency and route of administration of use and/or dosage may be considered by the QI on a case-by-case basis prior to recommending an appropriate washout or their enrollment in the study.

1. Oral NSAIDs or topical application on the target knee
2. Narcotics
3. Oral corticosteroids or topical application on the target knee
4. Oral analgesics except acetaminophen as a rescue medication or topical application on the target knee
5. Digoxin
6. Anti-hypertensive drugs
7. Anticoagulants or antiplatelet drugs
8. Medications used for OA treatment
9. Diazepam

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Change in knee joint function: Pain | 12 weeks
  This will be determined by change in pain of the identified knee joint from baseline to 12-week post-supplementation between JointAlive™ and placebo, as assessed by Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) pain and stiffness scores. Questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain. The lowest number represents no pain while the highest number represent extreme pain or stiffness. These are then converted to the Knee injury and Osteoarthritis Outcomes Score (KOOS) pain scores. KOOS scoring system ranges from 1-100, with 0 representing no pain and 100 being extreme pain.
Change in knee joint function: Stiffness | 12 weeks
  This will be determined by change in stiffness of the identified knee joint from baseline to 12-week post-supplementation between JointAlive™ and placebo, as assessed by Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) pain and stiffness scores. Questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible 0-8 for Stiffness. The lowest number represents no pain or stiffness while the highest number represent extreme pain or stiffness. These are then converted to the Knee injury and Osteoarthritis Outcomes Score (KOOS) pain scores. KOOS scoring system ranges from 1-100, with 0 representing no stiffness and 100 being extreme stiffness.

SECONDARY OUTCOMES:
Change in Pain | 6 weeks
  Change in pain of the identified knee joint from baseline to 6-week post-supplementation between JointAlive™ and placebo, as assessed by Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) pain and stiffness scores. Questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain. The lowest number represents no pain while the highest number represent extreme pain or stiffness. These are then converted to the Knee injury and Osteoarthritis Outcomes Score (KOOS) pain scores. KOOS scoring system ranges from 1-100, with 0 representing no pain and 100 being extreme pain.
Change in Stiffness | 6 weeks
  Change in stiffness of the identified knee joint from baseline to 6-week post-supplementation between JointAlive™ and placebo, as assessed by Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) pain and stiffness scores. Questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible 0-8 for Stiffness. The lowest number represents no pain or stiffness while the highest number represent extreme pain or stiffness. These are then converted to the Knee injury and Osteoarthritis Outcomes Score (KOOS) pain scores. KOOS scoring system ranges from 1-100, with 0 representing no stiffness and 100 being extreme stiffness.
Knee OA symptoms as assessed by KOOS symptoms score | 6-12 weeks
  KOOS Scores range from 0 to 100. A score of 0 indicates the worst possible knee symptoms and 100 indicates no knee symptoms.
Daily physical function as assessed by KOOS in function daily living score | 6-12 weeks
  The Scoring system ranges from 0 to 100, with 0 representing extreme problems and 100 representing no problems
Physical function in sports and recreational activities as assessed by KOOS function in sports and recreational activities score | 6-12 weeks
  The Scoring system ranges from 0 to 100, with 0 representing extreme problems with physical functions and 100 representing no problems
Current pain as assessed by Pain Visual Analogue Scale (VAS) scores | 6-12 weeks
  The Pain VAS questionnaire is a unidimensional measure of pain intensity. With the use of a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100 depending on pain intensity. A score of 0 represents no pain while a score of 100 represents extreme pain.
Quality of life as assessed by Short Form 36 (SF-36) Questionnaire and KOOS quality of life score | 6-12 weeks
  The Scoring system ranges from 0 to 100, with 0 representing poorest quality of life and 100 representing no problems
Knee joint range of motion (flexion and extension) as assessed by a knee goniometer | 6-12 weeks
Serum level of C reactive protein (CRP) | 6-12 weeks
Use of acetaminophen as a rescue medication as assessed by study diary | 6-12 weeks

OTHER OUTCOMES:
Incidence of pre-emergent and post-emergent adverse events | 12 weeks
Blood pressure (BP) | 12 weeks
  Diastolic and systolic blood pressure (BP) after 6 and 12 weeks of supplementation with JointAlive™
Heart Rate | 12 weeks
  Heart rate (HR) after 6 and 12 weeks of supplementation with JointAlive™
Change alanine aminotransferase (ALT) after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change aspartate aminotransferase (AST) after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change alkaline phosphatase (ALP), after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in total bilirubin after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in total creatinine after 12 weeks of supplementation with JointAlive™ compared to placebo | 12 weeks
Change in electrolytes (Na+, K+, Cl-) after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in estimated glomerular filtration rate (eGFR) after 12 weeks of supplementation with JointAlive™ compared to placebo | 12 weeks
Change in white blood cell (WBC) count after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in neutrophils after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in lymphocytes after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in monocytes after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in eosinophils after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in basophils after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in red blood cell (RBC) count after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in hemoglobin after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in hematocrit after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in platelet count after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in mean corpuscular volume (MCV) after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in mean corpuscular hemoglobin (MCH) after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in mean corpuscular hemoglobin concentration (MCHC) after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in red cell distribution width (RDW) after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks
Change in mean platelet volume (MPV) after 12 weeks of supplementation with JointAlive™ compared to placebo. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Helmick CG, Felson DT, Lawrence RC, Gabriel S, Hirsch R, Kwoh CK, Liang MH, Kremers HM, Mayes MD, Merkel PA, Pillemer SR, Reveille JD, Stone JH; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part I. Arthritis Rheum. 2008 Jan;58(1):15-25. doi: 10.1002/art.23177. PMID 18163481
- [Background] Wallace IJ, Worthington S, Felson DT, Jurmain RD, Wren KT, Maijanen H, Woods RJ, Lieberman DE. Knee osteoarthritis has doubled in prevalence since the mid-20th century. Proc Natl Acad Sci U S A. 2017 Aug 29;114(35):9332-9336. doi: 10.1073/pnas.1703856114. Epub 2017 Aug 14. PMID 28808025
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Litwic A, Edwards MH, Dennison EM, Cooper C. Epidemiology and burden of osteoarthritis. Br Med Bull. 2013;105:185-99. doi: 10.1093/bmb/lds038. Epub 2013 Jan 20. PMID 23337796
- [Background] Losina E, Paltiel AD, Weinstein AM, Yelin E, Hunter DJ, Chen SP, Klara K, Suter LG, Solomon DH, Burbine SA, Walensky RP, Katz JN. Lifetime medical costs of knee osteoarthritis management in the United States: impact of extending indications for total knee arthroplasty. Arthritis Care Res (Hoboken). 2015 Feb;67(2):203-15. doi: 10.1002/acr.22412. PMID 25048053
- [Background] Salmon JH, Rat AC, Sellam J, Michel M, Eschard JP, Guillemin F, Jolly D, Fautrel B. Economic impact of lower-limb osteoarthritis worldwide: a systematic review of cost-of-illness studies. Osteoarthritis Cartilage. 2016 Sep;24(9):1500-8. doi: 10.1016/j.joca.2016.03.012. Epub 2016 Mar 23. PMID 27034093
- [Background] Heidari B. Knee osteoarthritis prevalence, risk factors, pathogenesis and features: Part I. Caspian J Intern Med. 2011 Spring;2(2):205-12. PMID 24024017
- [Background] Chen D, Shen J, Zhao W, Wang T, Han L, Hamilton JL, Im HJ. Osteoarthritis: toward a comprehensive understanding of pathological mechanism. Bone Res. 2017 Jan 17;5:16044. doi: 10.1038/boneres.2016.44. eCollection 2017. PMID 28149655
- [Background] Kohn MD, Sassoon AA, Fernando ND. Classifications in Brief: Kellgren-Lawrence Classification of Osteoarthritis. Clin Orthop Relat Res. 2016 Aug;474(8):1886-93. doi: 10.1007/s11999-016-4732-4. Epub 2016 Feb 12. No abstract available. PMID 26872913
- [Background] Felson DT, Hodgson R. Identifying and treating preclinical and early osteoarthritis. Rheum Dis Clin North Am. 2014 Nov;40(4):699-710. doi: 10.1016/j.rdc.2014.07.012. Epub 2014 Sep 12. PMID 25437286
- [Background] Ayhan E, Kesmezacar H, Akgun I. Intraarticular injections (corticosteroid, hyaluronic acid, platelet rich plasma) for the knee osteoarthritis. World J Orthop. 2014 Jul 18;5(3):351-61. doi: 10.5312/wjo.v5.i3.351. eCollection 2014 Jul 18. PMID 25035839
- [Background] Charlesworth J, Fitzpatrick J, Perera NKP, Orchard J. Osteoarthritis- a systematic review of long-term safety implications for osteoarthritis of the knee. BMC Musculoskelet Disord. 2019 Apr 9;20(1):151. doi: 10.1186/s12891-019-2525-0. PMID 30961569
- [Background] Fang J, Zhang Y. Icariin, an Anti-atherosclerotic Drug from Chinese Medicinal Herb Horny Goat Weed. Front Pharmacol. 2017 Oct 12;8:734. doi: 10.3389/fphar.2017.00734. eCollection 2017. PMID 29075193
- [Background] Chen SR, Xu XZ, Wang YH, Chen JW, Xu SW, Gu LQ, Liu PQ. Icariin derivative inhibits inflammation through suppression of p38 mitogen-activated protein kinase and nuclear factor-kappaB pathways. Biol Pharm Bull. 2010;33(8):1307-13. doi: 10.1248/bpb.33.1307. PMID 20686223
- [Background] Liu MH, Sun JS, Tsai SW, Sheu SY, Chen MH. Icariin protects murine chondrocytes from lipopolysaccharide-induced inflammatory responses and extracellular matrix degradation. Nutr Res. 2010 Jan;30(1):57-65. doi: 10.1016/j.nutres.2009.10.020. PMID 20116661
- [Background] Zu Y, Mu Y, Li Q, Zhang ST, Yan HJ. Icariin alleviates osteoarthritis by inhibiting NLRP3-mediated pyroptosis. J Orthop Surg Res. 2019 Sep 11;14(1):307. doi: 10.1186/s13018-019-1307-6. PMID 31511005
- [Background] Yan N, Wen DS, Zhao YR, Xu SJ. Epimedium sagittatum inhibits TLR4/MD-2 mediated NF-kappaB signaling pathway with anti-inflammatory activity. BMC Complement Altern Med. 2018 Nov 13;18(1):303. doi: 10.1186/s12906-018-2363-x. PMID 30424767
- [Background] Wang P, Zhang F, He Q, Wang J, Shiu HT, Shu Y, Tsang WP, Liang S, Zhao K, Wan C. Flavonoid Compound Icariin Activates Hypoxia Inducible Factor-1alpha in Chondrocytes and Promotes Articular Cartilage Repair. PLoS One. 2016 Feb 3;11(2):e0148372. doi: 10.1371/journal.pone.0148372. eCollection 2016. PMID 26841115
- [Background] Pan L, Zhang Y, Chen N, Yang L. Icariin Regulates Cellular Functions and Gene Expression of Osteoarthritis Patient-Derived Human Fibroblast-Like Synoviocytes. Int J Mol Sci. 2017 Dec 8;18(12):2656. doi: 10.3390/ijms18122656. PMID 29292760
- [Background] Luo Y, Zhang Y, Huang Y. Icariin Reduces Cartilage Degeneration in a Mouse Model of Osteoarthritis and is Associated with the Changes in Expression of Indian Hedgehog and Parathyroid Hormone-Related Protein. Med Sci Monit. 2018 Sep 23;24:6695-6706. doi: 10.12659/MSM.910983. PMID 30244259
- [Background] Wang F, Shi L, Zhang Y, Wang K, Pei F, Zhu H, Shi Z, Tao T, Li Z, Zeng P, Wang X, Ji Q, Qin L, Xue Q. A Traditional Herbal Formula Xianlinggubao for Pain Control and Function Improvement in Patients with Knee and Hand Osteoarthritis: A Multicenter, Randomized, Open-Label, Controlled Trial. Evid Based Complement Alternat Med. 2018 Feb 12;2018:1827528. doi: 10.1155/2018/1827528. eCollection 2018. PMID 29619064
- [Background] Wang L, Ma R, Liu C, Liu H, Zhu R, Guo S, Tang M, Li Y, Niu J, Fu M, Gao S, Zhang D. Salvia miltiorrhiza: A Potential Red Light to the Development of Cardiovascular Diseases. Curr Pharm Des. 2017;23(7):1077-1097. doi: 10.2174/1381612822666161010105242. PMID 27748194
- [Background] Ma S, Zhang D, Lou H, Sun L, Ji J. Evaluation of the anti-inflammatory activities of tanshinones isolated from Salvia miltiorrhiza var. alba roots in THP-1 macrophages. J Ethnopharmacol. 2016 Jul 21;188:193-9. doi: 10.1016/j.jep.2016.05.018. Epub 2016 May 10. PMID 27178632
- [Background] Bai B, Li Y. Danshen prevents articular cartilage degeneration via antioxidation in rabbits with osteoarthritis. Osteoarthritis Cartilage. 2016 Mar;24(3):514-20. doi: 10.1016/j.joca.2015.10.004. Epub 2015 Oct 17. PMID 26485068
- [Background] Xu X, Lv H, Li X, Su H, Zhang X, Yang J. Danshen attenuates osteoarthritis-related cartilage degeneration through inhibition of NF-kappaB signaling pathway in vivo and in vitro. Biochem Cell Biol. 2017 Dec;95(6):644-651. doi: 10.1139/bcb-2017-0025. Epub 2017 Jun 29. PMID 28662337
- [Background] Xu X, Lv H, Li X, Su H, Zhang X, Yang J. Danshen attenuates cartilage injuries in osteoarthritis in vivo and in vitro by activating JAK2/STAT3 and AKT pathways. Exp Anim. 2018 May 10;67(2):127-137. doi: 10.1538/expanim.17-0062. Epub 2017 Oct 31. PMID 29093428
- [Background] Ren J, Fu L, Nile SH, Zhang J, Kai G. Salvia miltiorrhiza in Treating Cardiovascular Diseases: A Review on Its Pharmacological and Clinical Applications. Front Pharmacol. 2019 Jul 5;10:753. doi: 10.3389/fphar.2019.00753. eCollection 2019. PMID 31338034
- [Background] Ou-Yang SH, Jiang T, Zhu L, Yi T. Dioscorea nipponica Makino: a systematic review on its ethnobotany, phytochemical and pharmacological profiles. Chem Cent J. 2018 May 11;12(1):57. doi: 10.1186/s13065-018-0423-4. PMID 29748731
- [Background] Junchao Y, Zhen W, Yuan W, Liying X, Libin J, Yuanhong Z, Wei Z, Ruilin C, Lu Z. Anti- trachea inflammatory effects of diosgenin from Dioscorea nipponica through interactions with glucocorticoid receptor alpha. J Int Med Res. 2017 Feb;45(1):101-113. doi: 10.1177/0300060516676724. Epub 2016 Dec 7. PMID 27913746
- [Background] Zhao X, Yin L, Fang L, Xu L, Sun P, Xu M, Liu K, Peng J. Protective effects of dioscin against systemic inflammatory response syndromevia adjusting TLR2/MyD88/NF-kappab signal pathway. Int Immunopharmacol. 2018 Dec;65:458-469. doi: 10.1016/j.intimp.2018.10.036. Epub 2018 Oct 31. PMID 30390593
- [Background] Collins NJ, Prinsen CA, Christensen R, Bartels EM, Terwee CB, Roos EM. Knee Injury and Osteoarthritis Outcome Score (KOOS): systematic review and meta-analysis of measurement properties. Osteoarthritis Cartilage. 2016 Aug;24(8):1317-29. doi: 10.1016/j.joca.2016.03.010. Epub 2016 Mar 21. PMID 27012756
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558
- [Background] Rosemann T, Joos S, Koerner T, Szecsenyi J, Laux G. Comparison of AIMS2-SF, WOMAC, x-ray and a global physician assessment in order to approach quality of life in patients suffering from osteoarthritis. BMC Musculoskelet Disord. 2006 Jan 26;7:6. doi: 10.1186/1471-2474-7-6. PMID 16438717
- [Background] Berenbaum F, Grifka J, Brown JP, Zacher J, Moore A, Krammer G, Dutta D, Sloan VS. Efficacy of lumiracoxib in osteoarthritis: a review of nine studies. J Int Med Res. 2005 Jan-Feb;33(1):21-41. doi: 10.1177/147323000503300102. PMID 15651713
- [Background] Wessel J. The reliability and validity of pain threshold measurements in osteoarthritis of the knee. Scand J Rheumatol. 1995;24(4):238-42. doi: 10.3109/03009749509100881. PMID 7481589
- [Background] Escobar A, Quintana JM, Bilbao A, Arostegui I, Lafuente I, Vidaurreta I. Responsiveness and clinically important differences for the WOMAC and SF-36 after total knee replacement. Osteoarthritis Cartilage. 2007 Mar;15(3):273-80. doi: 10.1016/j.joca.2006.09.001. Epub 2006 Oct 17. PMID 17052924
- [Background] Giordano N, Fioravanti A, Papakostas P, Montella A, Giorgi G, Nuti R. The efficacy and tolerability of glucosamine sulfate in the treatment of knee osteoarthritis: A randomized, double-blind, placebo-controlled trial. Curr Ther Res Clin Exp. 2009 Jun;70(3):185-96. doi: 10.1016/j.curtheres.2009.05.004. PMID 24683229
- [Derived] Li L, Wang Y, Wang S, Zong J, Zhang Z, Zou S, Zhao Z, Cao Y, Liu Z. A Randomized, Double-Blind, Placebo-Controlled Study Investigating the Safety and Efficacy of a Herbal Formulation on Knee Joint Function in Adults with Knee Osteoarthritis. J Integr Complement Med. 2025 Jan;31(1):54-63. doi: 10.1089/jicm.2023.0124. Epub 2024 Oct 14. PMID 39400265
- See also: FDA Drug Safety Communication: FDA strengthens warning that non-aspirin nonsteroidal anti-inflammatory drugs (NSAIDs) can cause heart attacks or strokes — https://www.fda.gov/drugs/drug-safety-and-availability/fda-drug-safety-communication-fda-strengthens-warning-non-aspirin-nonsteroidal-anti-inflammatory
- See also: KOOS Scoring guide — http://www.koos.nu/